CLINICAL TRIAL: NCT06813482
Title: Heart Health at Home - Real-World Evaluation of a Digitally Enabled Cardiac Rehabilitation Program
Brief Title: Real-World Evaluation of a Digitally Enabled Cardiac Rehabilitation Program
Status: Completed | Type: Observational
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: University of Melbourne (Other); Medibank (Unknown)
Responsible Party: Sponsor
Other Study IDs: 321/21
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Heart Disease; Chronic Disease; Cardiovascular Disease Prevention
Keywords: telerehabilitation; cardiac rehabilitation; Digital health
MeSH Terms: conditions — Heart Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DeCR: Heart Health at Home - Digitally enabled cardiac rehabilitation
  Interventions: Behavioral: Digitally enabled cardiac rehabilitation
- F2F-CR: Traditional Face-to-Face Cardiac Rehabilitation
  Interventions: Behavioral: F2F-CR
- Usual Care: Usual Care - eligible for cardiac rehabilitation and who unlikely participated in any formal cardiac rehabilitation program
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Digitally enabled cardiac rehabilitation — The intervention consists of an 8-week remotely delivered cardiac rehabilitation program. It includes an initial assessment during week 1, six weeks of participation in a digitally enabled cardiac rehabilitation (DeCR) program (weeks 2-7), and a final assessment in week 8. Participants will utilize a digital mobile application and receive weekly telehealth consultations with a cardiac nurse. The program is designed to facilitate behavior change and improve outcomes through the following modalities:
  1. Telehealth - individualized coaching delivered via telephone by a cardiac nurse, to ensure that patient's take their medications as prescribed and to give health education and guidance on lifestyle changes.
  2. Mobile application (called SmartCR) and nurse web portal - for remote monitoring and personalized care planning. The app monitors health and physical activity, has prompted tasks and delivers education via video, audio and written articles.
  Groups: DeCR
Behavioral: F2F-CR — Traditional Face-to-face cardiac rehabilitation
  Groups: F2F-CR
Behavioral: Usual Care Group — Usual Care - eligible for cardiac rehabilitation and who unlikely participated in any formal cardiac rehabilitation program
  Groups: Usual Care

SUMMARY:
After a heart event or procedure, patients are encouraged to participate in a cardiac rehabilitation (CR) program to improve their health and reduce the risk of future problems. These programs have been shown to improve heart health and reduce hospital readmissions and deaths. However, many patients face challenges attending in-person CR programs, particularly those residing in regional or remote areas. As a result, many patients worldwide do not participate in CR.

Missing out on CR increases the risk of unplanned hospital visits. To overcome these challenges, digitally enabled cardiac rehabilitation programs provide an alternative. These programs use technology, such as mobile apps and telehealth, to deliver care remotely. Although these programs have the potential to make CR more accessible, there is still limited evidence about how well they work in real-world settings, including their impact on hospital visits and overall healthcare use.

Therefore, the goal of this real-world observational study is to evaluate if a digitally enabled and remotely delivered cardiac rehabilitation (DeCR) program, called Heart Health at Home, can improve risk factors and hospital utilization in adults who have experienced a heart event or undergone a heart procedure.

The questions it aims to answer are:

1. Does the DeCR intervention group have associated reductions in hospital readmissions, total hospital bed days, and mortality compared to the usual care group?
2. Do DeCR intervention patients have similar hospital utilization outcomes compared to traditional face-to-face cardiac rehabilitation patients?
3. Does the DeCR intervention have associated improvements in healthy lifestyle behaviors and clinical risk factors?
4. Does the DeCR intervention increase uptake and engagement to cardiac rehabilitation and what are participants' and cardiac nurses' experiences and perceptions of the program?
5. Is the DeCR intervention cost effective?

Researchers will compare participants receiving the DeCR intervention to those receiving traditional face-to-face cardiac rehabilitation and usual care to see if the program leads to better health outcomes and reduced healthcare utilization.

Participants will participate in an 8-week DeCR intervention entailing telehealth consultations with a cardiac rehabilitation nurse and they will use a mobile app, called SmartCR, to access education, remote monitoring and progress tracking.

DETAILED DESCRIPTION:
The Investigators aim to assess a digitally enabled cardiac rehabilitation (DeCR) program, called Heart Health at Home, implemented in a real-world setting. The investigators will assess whether the program improves clinical outcomes, healthcare utilization, and program engagement for adults recovering from a cardiac event or procedure. The researchers hypothesize that the intervention would be associated with healthy lifestyle changes and improvements in clinical risk factors. They anticipate that Heart Health at Home would be associated with similar outcomes compared to traditional face-to-face cardiac rehabilitation and reduced hospital readmissions, hospital bed days and mortality compared to usual care.

Methods:

Investigators will evaluate this study via a prospective cohort study, to establish the associated benefits of the program on healthy lifestyle changes and improvements in clinical risk factors, followed by a propensity matched cohort study via analysis of private hospital claims data. Using propensity score matching methods, two concurrent control groups will be established to compare the DeCR group with patients who undertook either: 1) Face-to-Face cardiac rehabilitation (F2F-CR) or 2) usual care, following an index cardiac hospitalization. The investigators will assess the associated outcomes of DeCR participation on recurrent hospitalisations, days spent in hospital, mortality and cost outlays within 12 months post index admission. Additionally, the investigators will examine participants' and cardiac nurses' experiences and perceptions of the DeCR program.

Patients aged over 18 years, who hold private health insurance with a large Australian private health insurer and who have been hospitalized with a cardiovascular diagnosis and/or procedure eligible for cardiac rehabilitation will be recruited. Patients will be excluded if they; 1) have heart failure (due to the potential for more specialized care); 2) are attending an alternate cardiac rehabilitation program and; 3) do not have access to a smart phone and internet connection.

Baseline pre vs post measures will include:

1. Self-reported demographic information (assessed prior to the intervention) - age, sex, ethnicity, employment, living situation, location and geographic based socioeconomic status.
2. Self reported risk factors - blood pressure using an automated device, height and weight, cigarette smoking, diet via a 9-item questionnaire developed by the investigators based on dietary guidelines, alcohol (total standard drinks per week) and physical activity (total minutes per week).
3. Self reported health and lifestyle behaviours - medication adherence via the 4-item Morisky Medication Adherence Scale (MMAS); functional capacity via the 12-item Duke Activity Status Index (DASI); psychological distress via the Kessler Psychological Distress Scale (K10); health status via the EuroQol 5-level questionnaire (EQ-5D-5L) (index value-Australia) and patient engagement in managing their health via the 13-item Patient Activation Measure (PAM).
4. App engagement tasks via the mobile app - daily blood pressure, using an automated device, stress levels, twice daily walking, weekly weight measurements and personalised education topics. Blood glucose concentration and alcohol intake will only be assessed if assigned to patients as a goal.

Hospital admission data will be collected for all patient groups, for 12-months post discharge and include:

date of admission and discharge, index procedure information, sociodemographic data, cardiovascular disease condition, smoking history, past history of diabetes, chronic kidney disease and previous acute myocardial infarction, Charlson Comorbidity Index and risk of readmission via the PEGASUS-TIMI score - 'Prevention with Ticagrelor of Secondary Thrombotic events in high-risk Patients with Prior Acute Coronary Syndrome - Thrombolysis in Myocardial Infarction'.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years AND
2. hold private health insurance with Medibank at a level that includes cover for hospital treatment AND
3. Discharged from hospital with a cardiovascular diagnosis and/or procedure eligible for cardiac rehabilitation, as defined by the National Heart Foundation of Australia AND
4. be able to give written consent to participate

Exclusion Criteria:

1. Patients with heart failure; OR
2. Patients attending an alternate cardiac rehab program for the corresponding index event; OR
3. Patients who do not have access to a smart phone and internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Privately insured Australian patients, residing in any State or Territory in Australia
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Hospital utilization | 30-day, 90-day and 12-month post discharge
  All cause rehospitalizations, and hospital bed-days
Hospital utilization | 30-day, 90-day and 12-month post discharge
  Cardiac related rehospitalizations, and hospital bed-days
Mortality | 30-days and 12-month post discharge
  All cause Mortality

SECONDARY OUTCOMES:
Blood pressure | At completion of the intervention at 8 weeks.
  Pre vs post change in systolic and diastolic blood pressure (mmHg)
Body mass index | At completion of the intervention at 8 weeks.
  Pre vs post change in body mass index (BMI)
Diet | At completion of the intervention at 8 weeks
  Pre vs post change in diet score (9-item questionnaire developed by the investigator working group based on dietary guidelines). Scores range from a lowest of 9 to a high of 28. Higher scores denote better diet quality.
Alcohol intake - average number of standard alcoholic drinks consumed per week | At completion of the intervention at 8 weeks
  Pre vs post change in the average number of standard alcoholic drinks consumed per week
Physical activity | At completion of the intervention at 8 weeks
  Pre vs post change in the average number of minutes of physical activity completed per week (minutes per week).
Patient Activation Measure | At completion of the intervention at 8 weeks
  Pre vs post change in the Patient Activation Measure (PAM), which measures the knowledge, skills and confidence that a person has to manage their own wellbeing. Validated questionnaire comprising 13 questions. Score ranges from 0 to 100 with a higher score indicating greater patient activation. The minimum score is 0 and the maximum score is 100.
Functional capacity - Duke Activity Status Index | At completion of the intervention at 8 weeks
  Pre vs post change in the Duke Activity Status Index (DASI). Responses are summed to get a total score, which ranges from 0 to 58.2. Higher scores indicate higher functional capacity.
Kessler Psychological Distress Scale | At completion of the intervention at 8 weeks.
  Pre vs post change in the Kessler Psychological Distress Scale (K10). Higher scores denote worse psychological distress. The maximum score is 50, indicating severe distress and the minimum score is 10, indicating no distress.
Quality of life - EuroQol-5 Dimension questionnaire | At completion of the intervention at 8 weeks.
  Pre vs post change in quality of life via the EQ-5D-5L index value-Australia. The maximum score represents "perfect health" and is denoted as "1", while the minimum score represents the worst possible health state and is "0".
Medication adherence - 4-item Morisky Medication Adherence Scale | At completion of the intervention at 8 weeks.
  Pre vs post change in the 4-item Morisky Medication Adherence Scale (MMAS). The maximum score is 4 and the minimum score is 0. A higher score indicates better adherence, while a lower score suggests poorer adherence.

OTHER OUTCOMES:
Mobile app engagement for tasks set | At completion of the intervention at 8 weeks.
  Patient engagement for tasks set within the SmartCR app to be calculated by the number of tasks marked as completed, divided by the number of tasks assigned during the intervention period
Medication engagement via the app | At completion of the intervention at 8 weeks.
  Medication engagement via the app will be calculated by the number of medication reminders marked as taken or not taken, divided by the total number of medication reminders sent over the intervention period
Overall mobile app engagement | At completion of the intervention at 8 weeks.
  A composite variable to assess overall app engagement will be created by combining responses to tasks assigned and medication reminders.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda J Carrington, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
After de-identification and underlying published results, the data underlying the study may be shared on reasonable request to the Principal Investigator and approval by the Contributors. The deidentified data may only be available to researchers who provide a methodologically sound proposal, case-by-case basis at the discretion of Principal Investigator and study Contributors.
Time Frame: Following publication; no end date
Access Criteria: Access subject to approvals by Principal Investigator and study Contributors
URL: http://baker.edu.au/research/laboratories/preclinical-disease-prevention

REFERENCES:
- [Background] Blacher J, Olie V, Gabet A, Cinaud A, Tuppin P, Iliou MC, Grave C. Two-year prognosis and cardiovascular disease prevention after acute coronary syndrome: the role of cardiac rehabilitation-a French nationwide study. Eur J Prev Cardiol. 2024 Nov 18;31(16):1939-1947. doi: 10.1093/eurjpc/zwae194. PMID 38832727
- [Background] Kotseva K, Wood D, De Bacquer D; EUROASPIRE investigators. Determinants of participation and risk factor control according to attendance in cardiac rehabilitation programmes in coronary patients in Europe: EUROASPIRE IV survey. Eur J Prev Cardiol. 2018 Aug;25(12):1242-1251. doi: 10.1177/2047487318781359. Epub 2018 Jun 6. PMID 29873511
- [Background] Ades PA, Keteyian SJ, Wright JS, Hamm LF, Lui K, Newlin K, Shepard DS, Thomas RJ. Increasing Cardiac Rehabilitation Participation From 20% to 70%: A Road Map From the Million Hearts Cardiac Rehabilitation Collaborative. Mayo Clin Proc. 2017 Feb;92(2):234-242. doi: 10.1016/j.mayocp.2016.10.014. Epub 2016 Nov 15. PMID 27855953
- [Background] Woodruffe S, Neubeck L, Clark RA, Gray K, Ferry C, Finan J, Sanderson S, Briffa TG. Australian Cardiovascular Health and Rehabilitation Association (ACRA) core components of cardiovascular disease secondary prevention and cardiac rehabilitation 2014. Heart Lung Circ. 2015 May;24(5):430-41. doi: 10.1016/j.hlc.2014.12.008. Epub 2015 Jan 12. PMID 25637253
- [Background] Braver J, Marwick TH, Oldenburg B, Issaka A, Carrington MJ. Digital Health Programs to Reduce Readmissions in Coronary Artery Disease: A Systematic Review and Meta-Analysis. JACC Adv. 2023 Sep 7;2(8):100591. doi: 10.1016/j.jacadv.2023.100591. eCollection 2023 Oct. PMID 38938339
- [Background] Varnfield M, Karunanithi M, Lee CK, Honeyman E, Arnold D, Ding H, Smith C, Walters DL. Smartphone-based home care model improved use of cardiac rehabilitation in postmyocardial infarction patients: results from a randomised controlled trial. Heart. 2014 Nov;100(22):1770-9. doi: 10.1136/heartjnl-2014-305783. Epub 2014 Jun 27. PMID 24973083
- [Background] Golbus JR, Lopez-Jimenez F, Barac A, Cornwell WK 3rd, Dunn P, Forman DE, Martin SS, Schorr EN, Supervia M; Exercise, Cardiac Rehabilitation and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Quality of Care and Outcomes Research; and Council on Cardiovascular and Stroke Nursing. Digital Technologies in Cardiac Rehabilitation: A Science Advisory From the American Heart Association. Circulation. 2023 Jul 4;148(1):95-107. doi: 10.1161/CIR.0000000000001150. Epub 2023 Jun 5. PMID 37272365
- [Background] Turk-Adawi K, Sarrafzadegan N, Grace SL. Global availability of cardiac rehabilitation. Nat Rev Cardiol. 2014 Oct;11(10):586-96. doi: 10.1038/nrcardio.2014.98. Epub 2014 Jul 15. PMID 25027487
- [Background] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- See also: Baker Institute study website — https://baker.edu.au/research/laboratories/community-prevention-cardiac-research/project-medibank-heart-study